CLINICAL TRIAL: NCT07252934
Title: Enhancing District Health Centre Membership Among Older Adults Through Intergenerational Home-based and AI-generated Digital Interventions
Brief Title: District Health Centre Membership Among Older Adults in Hong Kong
Acronym: DHCRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wanjia, Aaron HE, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHCRCT
Record Dates: First submitted 2025-09-25; First posted 2025-11-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education on primary health care utilization (Experimental): Participants will receive education on primary healthcare services and their benefits for improving health outcomes. The education program includes a 1.5-hour face-to-face, home-based session and a 4-week AI-generated digital intervention.
  Interventions: Behavioral: Home-based and AI-generated digital intervention
- Education on general health (Active Comparator): Participants will receive general health education relevant to older adults. The program also includes a 1.5-hour face-to-face, home-based session and a 4-week AI-generated digital intervention.
  Interventions: Behavioral: Home-based and AI-generated digital intervention

INTERVENTIONS:
Behavioral: Home-based and AI-generated digital intervention — The home-based intervention is a 90-minute face-to-face session, during which trained student interns collect health assessment data and deliver theme-based, tailored health interventions. The digital intervention is a 1-month follow-up support involving daily messages via instant messaging apps (e.g., WhatsApp) that include health-related infographics, videos, and personalized advice.

SUMMARY:
This study is a cluster randomized controlled trial study to evaluate the feasibility, acceptability, and effectiveness of intergenerational home-based and AI-generated digital interventions in improving the proportion of District Health Centre members among older adults in Hong Kong.

DETAILED DESCRIPTION:
This is a two-group parallel cluster randomized controlled trial, involving 180 older adults recruited from 6 clusters. Clusters would be allocated to either the intervention or control arm in a 1:1 ratio Participants will receive home-based DHC intervention by trained students, followed by 1-month of AI-generated digital interventions, including infographics, videos, and messages on the introduction and promotion of DHC, via WhatsApp. The primary outcome is to increase the proportion of District Health Centre members. Secondary outcomes include the proportion of participants utilizing DHC services, physical well-being, mental health, and feasibility metrics. Data will be collected via surveys at baseline and follow-ups (1, 3, and 6 months).

This proposed pilot study aims to improve primary healthcare service uptake among older adults in Hong Kong. In doing so, it seeks to support healthier aging, improve health outcomes, alleviate pressure on hospitals, and offer evidence-based framework for addressing the needs of aging populations.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* spoke Chinese
* are physically, mentally, and cognitively capable of engaging in simple physical tasks
* understanding survey questions
* non district health centre member

Exclusion Criteria:

* All subjects have the right to withdraw if they wish not to continue

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
District health centre membership | 3 months
  The primary outcome is the proportion of older adults who become DHC members at 3 months.

SECONDARY OUTCOMES:
District health centre utilization | 3 months
  The proportion of older adults utilizing DHC service after 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He AWJ, Yuan R, Luk TT, Wang KMP, Chan SSC. Boosting Digital Health Engagement Among Older Adults in Hong Kong: Pilot Pre-Post Study of the Generations Connect Project. JMIR Form Res. 2025 May 8;9:e69611. doi: 10.2196/69611. PMID 40340793
- [Background] Wan Jia Aaron H, Yuan R, Chan SCS. Socio-demographic and behavioral predictors of multiple-dose COVID-19 vaccine uptake among older adults in Hong Kong: A community-based cross-sectional study of the generations connect project. Vaccine. 2025 Aug 13;61:127308. doi: 10.1016/j.vaccine.2025.127308. Epub 2025 Jun 2. PMID 40460652